CLINICAL TRIAL: NCT01817959
Title: A Phase 3, Multicenter, Randomized, Double-blind, Parallel Assignment Study to Assess the Efficacy and Safety of Reparixin in Pancreatic Islet Transplantation
Brief Title: Study to Assess Efficacy & Safety of Reparixin in Pancreatic Islet Transplantation
Acronym: REP0211
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REP0211; 2011-006201-10 (EudraCT Number)
Record Dates: First submitted 2013-03-07; First posted 2013-03-26 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2021-09

CONDITIONS: Islet Transplantation in Diabetes Mellitus Type 1
Keywords: Pancreatic islet transplantation; Diabetes Mellitus Type 1; Islet transplantation graft survival & function
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — reparixin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reparixin group (Experimental): Continuous iv infusion
  Interventions: Drug: Reparixin
- Placebo group (Placebo Comparator): Continuous iv infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Reparixin — Continuous i.v. infusion into a central vein for 7 days, starting approximately 12 hrs (6-18 hrs) before each pancreatic islet infusion.The Investigational Product (IP) were to be administered as an add-on treatment for the immunosuppressant regimen.
  Other Names: REP
  Arms: Reparixin group
Drug: Placebo — Continuous infusion at a volume/rate matching active treatment.The placebo was to be administered as well as an add-on treatment for the immunosuppressant regimen.
  Arms: Placebo group

SUMMARY:
The objective of this clinical trial was:

- to assess whether Reparixin leads to improved transplant outcome as measured by glycaemic control following intra-hepatic infusion of pancreatic islets in patients with Type 1 diabetes (T1D). The safety of Reparixin in the specific clinical setting was also evaluated.

Background: The chemokine CXCL8 plays a key role in the recruitment and activation of polymorphonuclear neutrophils in post-ischemia reperfusion injury after organ transplantation. Reparixin is the first low molecular weight blocker of CXCL8 biological activity in clinical development. Thus, the use of reparixin may emerge as a potential key component in the sequentially integrated approach to immunomodulation and control of non specific inflammatory events surrounding the early phases of pancreatic islet transplantation in T1D patients.

DETAILED DESCRIPTION:
Pancreatic islet transplantation has become a feasible option in the treatment of T1D which offers advantages over whole pancreas transplantation.

Several strategies are being evaluated, including anti-TNFα, aimed to prevent early inflammatory events that limit islet engraftment. Among possible mechanisms CXCL8 could play a crucial role in triggering the inflammatory reaction and might represent a relevant therapeutic target to prevent early graft failure.

Preliminary data obtained in transplanted patients recruited in the ongoing pilot trial coupled with the safety shown in human phase 1 and 2 studies provide a sound rationale for further development of reparixin in islet transplantation and prompted the conduct of this phase 3 clinical, multicentre, randomised, double-blind, parallel assignment study aimed at assessing the efficacy and safety of reparixin in preventing graft dysfunction after islet transplantation in T1D subjects.

At least 42 patients receiving pancreatic islet transplant were involved. Patients might receive up to 2 islet transplants, with the second transplant on average 6 months after the first one. Patients were randomly (2:1) assigned to receive either reparixin or placebo (control group). The Investigational Product was administered as an added on treatment to the immunosuppressant regimen.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years, inclusive.
* Patients eligible for a pancreatic islet transplantation program
* Planned intrahepatic islet transplantation alone from a non-living donor with brain death.
* Patients willing and able to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations.
* Patients who have given written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.

Exclusion Criteria:

* Recipients of any previous transplant, including recipients of previous pancreatic islet transplantation.
* Recipients of islet from a non-heart beating donor.
* Pre-transplant average daily insulin requirement >1 IU/kg/day.
* Pre-transplant (the more recent value obtained within the 4 months prior to enrolment) HbA1c >11%.
* Patients with inadequate renal reserve as per calculated creatinine clearance (CLcr) < 60 mL/min according to the Cockcroft-Gault formula (1976).
* Patients with hepatic dysfunction as defined by increased ALT (alanine aminotranferase) / AST (aspartate aminotransferase) > 3 x upper limit of normal (ULN) and increased total bilirubin > 3mg/dL [>51.3 µmol/L]).
* Patients who receive treatment for a medical condition requiring chronic use of systemic steroids.
* Treatment with any anti-diabetic medication other than insulin within 4 weeks of transplant.
* Use of any investigational agent within 12 weeks of enrolment, including "anti-inflammatory" strategies (e.g. anti-TNFα, anti-IL-1 RA).
* Hypersensitivity to:

  1. ibuprofen or to more than one non steroidal anti-inflammatory drug (NSAID).
  2. medications belonging to the class of sulfonamides, such as sulfamethazine, sulfamethoxazole, sulfasalazine, nimesulide or celecoxib.
* Pregnant or breast-feeding women; unwillingness to use effective contraceptive measures (females and males).

Additional exclusion criteria specific for US centre.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-10; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo PIEMONTI, MD, Principal Investigator — Dipartimento di Medicina Interna e Specialistica; IRCCS Ospedale San Raffaele; Torbjörn LUNDGREN, MD, PhD, Principal Investigator — Department of Transplantation Surgery; The Karolinska University Hospital; Gunnar TUFVESON, Professor, Principal Investigator — Department of Surgery; Uppsala University Hospital; Ehab RAFAEL, MD, PhD, Principal Investigator — Department of Nephrology and Transplantation; Skane University Hospital; James SHAW, Professor, Principal Investigator — Institute of Transplantation, Newcastle upon Tyne Hospitals - Freeman Hospital; Frantisek SAUDEK, MD, DrSc, Principal Investigator — Institute for Clinical and Experimental Medicine (IKEM), Department of Diabetes.; Piotr WITKOWSKI, MD, PhD, Principal Investigator — The University of Chicago Medical Center, Department of Surgery; Federico BERTUZZI, MD, Principal Investigator — S.S.D. Diabetologia, Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milano; Bengt GUSTAFSSON, MD, PhD, Principal Investigator — Transplant Institute - Sahlgrenska University Hospital
Locations (9):
- The University of Chicago Medical Center, Department of Surgery, Division of Abdominal Organ Transplantation, Chicago, Illinois, United States
- Institute for Clinical and Experimental Medicine (IKEM), Diabetes Centre; Department of Diabetes., Prague, Czechia
- Italy (2):
  - Dipartimento di Medicina Interna e Specialistica; IRCCS Ospedale San Raffaele, Milan
  - S.S.D. Diabetologia, Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Piazza Ospedale Maggiore 3, Milan
- Sweden (4):
  - Transplant Institute - Sahlgrenska University Hospital, Gothenburg
  - Department of Nephrology and Transplantation; Skane University Hospital, Malmo
  - Department of Transplantation Surgery; The Karolinska University Hospital, Stockholm
  - Division for Transplantation and Liver Surgery; Department of Surgery; Uppsala University Hospital, Uppsala
- Institute of Transplantation, Newcastle upon Tyne Hospitals - NHS Foundation Trust, Freeman Hospital, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Ajmal N, Bogart MC, Khan P, Max-Harry IM, Healy AM, Nunemaker CS. Identifying Promising Immunomodulators for Type 1 Diabetes (T1D) and Islet Transplantation. J Diabetes Res. 2024 Dec 20;2024:5151171. doi: 10.1155/jdr/5151171. eCollection 2024. PMID 39735417
- [Derived] Bachul PJ, Golab K, Basto L, Zangan S, Pyda JS, Perez-Gutierrez A, Borek P, Wang LJ, Tibudan M, Tran DK, Anteby R, Generette GS, Chrzanowski J, Fendler W, Perea L, Jayant K, Lucander A, Thomas C, Philipson L, Millis JM, Fung J, Witkowski P. Post-Hoc Analysis of a Randomized, Double Blind, Prospective Study at the University of Chicago: Additional Standardizations of Trial Protocol are Needed to Evaluate the Effect of a CXCR1/2 Inhibitor in Islet Allotransplantation. Cell Transplant. 2021 Jan-Dec;30:9636897211001774. doi: 10.1177/09636897211001774. PMID 33908301
- [Derived] Maffi P, Lundgren T, Tufveson G, Rafael E, Shaw JAM, Liew A, Saudek F, Witkowski P, Golab K, Bertuzzi F, Gustafsson B, Daffonchio L, Ruffini PA, Piemonti L; REP0211 Study Group. Targeting CXCR1/2 Does Not Improve Insulin Secretion After Pancreatic Islet Transplantation: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Trial in Type 1 Diabetes. Diabetes Care. 2020 Apr;43(4):710-718. doi: 10.2337/dc19-1480. Epub 2020 Feb 4. PMID 32019854

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 51 subjects were randomised into the trial. Three of these subjects did not have a transplant and never received randomised medication. Hence, a total of 48 subjects took trial medication and were included in the Safety Population.
Period: Overall Study
Arm/Group | Reparixin Group | Placebo Group
Started | 29 | 19
Completed | 25 | 16
Not Completed | 4 | 3
Not completed — Graft loss | 1 | 1
Not completed — forbidden medication | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Patient didn't proceed to 1st Islet Inf | 1 | 1

BASELINE CHARACTERISTICS:
Population: safety population: A total of 48 subjects (29 Reparixin, 19 placebo) received trial medication and therefore were included in the Safety Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Reparixin Group | Placebo Group | Total
Number analyzed (Participants) | 29 | 19 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 18 | 46
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (11.3) | 42.6 (10.8) | 45.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 12 | 7 | 19
Region of Enrollment [Number; unit: participants]
  Sweden | 7 | 6 | 13
  Czechia | 5 | 3 | 8
  United States | 8 | 4 | 12
  Italy | 7 | 5 | 12
  United Kingdom | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for the Serum C-peptide Level During the First 2 Hours of an MMTT (Mixed Meal Tolerance Test), Normalized by the Number of Islet Equivalent (IEQ)/kg
Description: The MMTT was to be performed ideally after an overnight fast. The test was to be initiated before 10 a.m. The Boost Original complete nutritional drink (Nestlé Nutrition) was used for the MMTT. Subjects were given 6 mL/kg of Boost preparation up to a maximum of 360 mL, to be drunk within 5 min. Blood samples for the C-peptide assay (the primary assessment) were withdrawn in fasting condition (basal), just prior to the meal (time 0, within 15 min prior to the meal) and then at 15, 30, 60, 90, 120 min after the meal.
Time Frame: Basal, -15' prior to meal, 15', 30', 60', 90', 120' following meal, Day 75±5 after the 1st islet infusion
Population: The Efficacy Population 1 consisted of all subjects who were randomised, received the IP (either Reparixin or placebo), and had a transplant (either one or two).
Measure: Mean (Standard Deviation); unit: ng/mL/min
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
ng/mL/min | 0.247 (0.218) | 0.321 (0.208)
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; Test type: Superiority; p = 0.9863, ANOVA — Treatment p value; least square mean difference = 0.001, 99.75% CI 2-sided [-0.205 to 0.207]

2. Primary Outcome: Area Under the Curve (AUC) for the Serum C-peptide Level During the First 2 Hours of an MMTT (Mixed Meal Tolerance Test), Normalized by the Number of Islet Equivalent (IEQ)/kg
Description: as for outcome 1
Time Frame: Basal, -15' prior to meal, 15', 30', 60', 90', 120' following meal, Day 365±14 after the last islet infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL/min
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 24 | 15
ng/mL/min | 0.234 (0.243) | 0.207 (0.127)
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; Test type: Superiority; p = 0.7115, ANOVA — Treatment p value; least square mean difference = 0.024, 99.75% CI 2-sided [-0.184 to 0.232]

3. Secondary Outcome: Percentage of Insulin-independent Patients at Day 75
Description: For the purpose of this study, insulin-independence is defined as freedom from the need to take exogenous insulin for 14 or more consecutive days, with adequate glycaemic control, as defined by:
  * a glycated hemoglobin (HbA1c) level of less than 7%;
  * a glucose level after an overnight fast not exceeding 140 mg/dL (7.8 mmol/L) more than three times a week (based on measuring capillary glucose level a minimum of 7 times in a 7 day period);
  * a glucose level not exceeding 2-hour postprandial levels of 180 mg/dL (10 mmol/L) more than four times a week (based on measuring capillary glucose level 14 times in a 7 day period).
Time Frame: Day 75±5 after the 1st and 2nd islet infusion
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
Percentage of participants
  transplant 1 | 18.5 | 5.6
  transplant 2: number analyzed (Participants) | 18 | 15
  transplant 2 | 27.8 | 53.3
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; Analytical statistics are reported for Day 75 after transplant 2; Test type: Superiority; p = 0.1346, Regression, Logistic — Treatment p value; Odds Ratio, log = 0.21, 95% CI 2-sided [0.03 to 1.63]

4. Secondary Outcome: Percentage of Insulin-independent Patients at Day 365
Description: as for outcome 3
Time Frame: Day 365±14 after last islet infusion
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 25 | 16
percentage of participants | 32.0 | 31.3
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; Test type: Superiority; p = 0.9130, Regression, Logistic — Treatment p value; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.17 to 4.93]

5. Secondary Outcome: Percentage of Patients Who Achieve and Maintain an HbA1c <7.0% (or a Reduction in HbA1c > 2%) AND Are Free of Severe Hypoglycaemic Events After Transplant in the Efficacy Population 1
Description: For the purpose of this study, a severe hypoglycaemic event is defined as an event with one of the following symptoms: memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness or visual symptoms, in which the subject was unable to treat him/herself and which was associated with either a blood glucose level <54mg/dL (3.0 mmol/L) or prompt recovery after oral carbohydrate, i.v. glucose, or glucagon administration.
Time Frame: HbA1c at Day 365±14 after the last islet infusion; severe hypoglycaemic events from Day 75 to Day 365 after the last islet infusion
Population: The Efficacy Population 1 consisted of all subjects who were randomised, received the IP (either Reparixin or placebo), and had a transplant (one or two).
Measure: Number; unit: Percentage of participants
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
Percentage of participants | 40.0 | 50.0
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; Test type: Superiority; p = 0.5467, Regression, Logistic — Treatment p value; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.16 to 2.66]

6. Secondary Outcome: Percentage of Patients Who Did Not Receive a 2nd Islet Infusion
Description: This endpoint describes subjects who were not allocated to a 2nd islet infusion because they were insulin independent after the 1st islet infusion.
Time Frame: Day 365±14 after the 1st islet infusion
Population: Efficacy Population 1 consisted of all subjects who were randomised, received the IP (either Reparixin or placebo), and had a transplant (either one or two).
Measure: Number; unit: percentage of participants
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
percentage of participants | 14.8 | 0.0
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; Test type: Superiority; p = 0.1383, Fisher Exact

7. Secondary Outcome: Cumulative Number of Severe Hypoglycaemic Events in the Efficacy Population 1
Description: The cumulative number of severe hypoglycaemic events after last transplant was assessed. For the purpose of this study, a severe hypoglycaemic event is defined as an event with one of the following symptoms: memory loss, confusion, uncontrollable behaviour, irrational behaviour, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness or visual symptoms, in which the subject was unable to treat him/herself and which was associated with either a blood glucose level <54 mg/dL (3.0 mmol/L) or prompt recovery after oral carbohydrate, i.v. glucose, or glucagon administration.
Time Frame: Day 365±14 after the last islet infusion
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 25 | 16
number of events | 2.88 (8.23) | 3.50 (7.65)

8. Secondary Outcome: Absolute Change From Baseline in Average Daily Insulin Requirements in Efficacy Population 1
Description: Change from baseline is assessed as absolute decrease from pre-transplant levels. For the purpose of this study, daily insulin is averaged over the previous week.
Time Frame: Day 75±5 after the 1st and 2nd islet infusion and day 365±14 after last islet infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
IU/kg/day
  transplant 1 | -0.231 (0.204) | -0.220 (0.203)
  transplant 2: number analyzed (Participants) | 18 | 15
  transplant 2 | -0.389 (0.163) | -0.463 (0.168)
  last transplant: number analyzed (Participants) | 25 | 16
  last transplant | -0.302 (0.167) | -0.375 (0.208)
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; This is is the analytic statistics for Day 75 (Transplant 1); Test type: Superiority; p = 0.6952, ANCOVA — Treatment p value; least square mean difference = -0.021, 95% CI 2-sided [-0.130 to 0.088]
Statistical Analysis 2: Comparison: Reparixin Group vs Placebo Group; This is is the analytic statistics for Day 75 (Transplant 2); Test type: Superiority; p = 0.5560, ANCOVA — This is a treatment p value; least square mean difference = 0.028, 95% CI 2-sided [-0.068 to 0.124]
Statistical Analysis 3: Comparison: Reparixin Group vs Placebo Group; This is the analytic statics for Day 365 (last Transplant); Test type: Superiority; p = 0.2537, ANCOVA — Treatment p value; Treatment p value; least square mean difference = 0.056, 95% CI 2-sided [-0.042 to 0.154]

9. Secondary Outcome: Percent Change From Baseline in Average Daily Insulin Requirements in Efficacy Population 1
Description: Change from baseline is assessed as percentage decrease from pre-transplant levels. For the purpose of this study, daily insulin is averaged over the previous week.
Time Frame: Day 75±5 after the 1st and 2nd islet infusion and day 365±14 after last islet infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
Percentage change
  Transplant 1 | -42.5 (54.1) | -35.0 (35.3)
  Transplant 2: number analyzed (Participants) | 18 | 15
  Transplant 2 | -74.0 (28.6) | -27.7 (26.3)
  Last transplant: number analyzed (Participants) | 25 | 16
  Last transplant | -59.4 (35.8) | -63.7 (33.7)
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; This is the analytic statics for Day 75 (Transplant 1); Test type: Superiority; p = 0.5910, ANCOVA — Treatment p value; least square mean difference = -7.4, 95% CI 2-sided [-35.2 to 20.3]
Statistical Analysis 2: Comparison: Reparixin Group vs Placebo Group; This is the analytic statics for Day 75 (Transplant 2); Test type: Superiority; p = 0.5966, ANCOVA — Treatment p value; Treatment p value; least square mean difference = 4.2, 95% CI 2-sided [-11.8 to 20.2]
Statistical Analysis 3: Comparison: Reparixin Group vs Placebo Group; This is the analytic statics for Day 365 (last Transplant); Test type: Superiority; p = 0.5005, ANCOVA — Treatment p value; least square mean difference = 6.1, 95% CI 2-sided [-12.1 to 24.4]

10. Secondary Outcome: Absolute Change in HbA1c % From Pre-transplant Levels in Efficacy Population 1
Description: Change from baseline in Glycated haemoglobin (HbA1c) was assessed as absolute decrease from pre-transplant levels. Diagnostic standards for HbA1c from American Diabetes Association are: <5.7% Normal; 5.7-6.4% prediabetes; >6.5 diabetes.
Time Frame: Day 75±5 after the 1st and 2nd islet infusion and day 365±14 after last islet infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of HbA1c
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
percent of HbA1c
  Transplant 1 | -1.58 (0.87) | -2.18 (1.23)
  Transplant 2: number analyzed (Participants) | 18 | 15
  Transplant 2 | -2.04 (1.10) | -2.81 (1.37)
  Last Transplant | -1.30 (1.14) | -1.87 (1.26)
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; This is the analytic statics for Day 75 (Transplant 1); Test type: Superiority; p = 0.3253, ANCOVA — Treatment p value; least square mean difference = 0.21, 95% CI 2-sided [-0.21 to 0.63]
Statistical Analysis 2: Comparison: Reparixin Group vs Placebo Group; This is the analytic statics for Day 75 (Transplant 2); Test type: Superiority; p = 0.6069, least square mean difference — Treatment p value; least square mean difference = 0.16, 95% CI 2-sided [-0.46 to 0.78]
Statistical Analysis 3: Comparison: Reparixin Group vs Placebo Group; This is the analytic statics for Day 365 (last Transplant); Test type: Superiority; p = 0.6437, ANCOVA — Treatment p value; Treatment p value; Least square mean difference = 0.17, 95% CI 2-sided [-0.56 to 0.93]

11. Secondary Outcome: Percent Change in HbA1c % From Pre-transplant Levels in Efficacy Population 1
Description: Change from baseline in Glycated haemoglobin (HbA1c) was assessed as percentage decrease from pre-transplant levels. Diagnostic standards for HbA1c from American Diabetes Association are: <5.7% Normal; 5.7-6.4% prediabetes; >6.5 diabetes.
Time Frame: Day 75±5 after the 1st and 2nd islet infusion and day 365+14 after last islet infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change of Hb1Ac %
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
Percent change of Hb1Ac %
  Transplant 1 | -18.9 (9.5) | -24.0 (10.6)
  Transplant 2: number analyzed (Participants) | 18 | 15
  Transplant 2 | -24.4 (11.6) | -30.5 (11.7)
  Last Transplant: number analyzed (Participants) | 25 | 16
  Last Transplant | -15.7 (13.1) | -20.9 (12.9)
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; This is the analytic statistics for Day 75 (Transplant 1); Test type: Superiority; p = 0.4290, ANCOVA — Treatment p value; least square mean difference = 2.0, 95% CI 2-sided [-3.0 to 6.9]
Statistical Analysis 2: Comparison: Reparixin Group vs Placebo Group; This is the analytic statistics for Day 75 (Transplant 2); Test type: Superiority; p = 0.7853, ANCOVA — Treatment p value; least square mean difference = 1.0, 95% CI 2-sided [-6.3 to 8.3]
Statistical Analysis 3: Comparison: Reparixin Group vs Placebo Group; This is the analytic statistics for Day 365 (last Transplant); Test type: Superiority; p = 0.6583, ANCOVA — Treatment p value; least square mean difference = 1.9, 95% CI 2-sided [-6.6 to 10.4]

12. Secondary Outcome: Basal (Fasting) and 0 to 120 Min Time Course of Glucose Derived From the Mixed Meal Tolerance Test (MMTT) in Efficacy Population 1
Description: Glucose levels were measured at the baseline in fasting condition, and at the following timepoints: 15, 30, 60, 90, 120 min after mixed meal at the hereunder reported time frame.
Time Frame: Day 75±5 after the 1st and 2nd islet infusion and day 365±14 after last islet infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
mg/dL
  Basal - day 75 - Transplant 1 | 120.6 (51.7) | 118.9 (40.2)
  15 min - day 75 - Transplant 1: number analyzed (Participants) | 26 | 17
  15 min - day 75 - Transplant 1 | 146.0 (56.0) | 132.5 (27.6)
  30 min - day 75 - Transplant 1: number analyzed (Participants) | 27 | 17
  30 min - day 75 - Transplant 1 | 191.6 (66.6) | 168.1 (50.0)
  60 min - day 75 - Transplant 1: number analyzed (Participants) | 27 | 17
  60 min - day 75 - Transplant 1 | 236.9 (86.0) | 219.1 (65.9)
  90 min - day 75 - Transplant 1: number analyzed (Participants) | 27 | 17
  90 min - day 75 - Transplant 1 | 254.0 (110.1) | 245.0 (84.7)
  120 min - day 75 - Transplant 1: number analyzed (Participants) | 27 | 16
  120 min - day 75 - Transplant 1 | 264.1 (116.7) | 246.0 (84.4)
  Basal - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  Basal - day 75 - Transplant 2 | 103.8 (19.8) | 112.8 (18.6)
  15 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  15 min - day 75 - Transplant 2 | 130.0 (22.3) | 134.8 (26.8)
  30 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  30 min - day 75 - Transplant 2 | 166.7 (33.6) | 157.8 (32.6)
  60 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  60 min - day 75 - Transplant 2 | 189.1 (57.9) | 172.0 (70.9)
  90 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  90 min - day 75 - Transplant 2 | 191.8 (72.8) | 175.1 (99.7)
  120 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  120 min - day 75 - Transplant 2 | 188.0 (88.1) | 171.7 (104.8)
  Basal - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  Basal - day 365 - Last transplant | 112.2 (37.6) | 125.1 (64.5)
  15 min - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  15 min - day 365 - Last transplant | 139.5 (43.1) | 146.7 (68.9)
  30 min - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  30 min - day 365 - Last transplant | 180.1 (53.9) | 182.7 (80.2)
  60 min - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  60 min - day 365 - Last transplant | 221.2 (81.2) | 213.6 (106.2)
  90 min - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  90 min - day 365 - Last transplant | 235.7 (112.6) | 222.0 (122.6)
  120 min - day 365 - Transplant 2: number analyzed (Participants) | 23 | 14
  120 min - day 365 - Transplant 2 | 239.9 (127.6) | 205.5 (104.3)

13. Secondary Outcome: Basal (Fasting) and 0 to 120 Min Time Course of C-peptide (Non-normalized) Derived From the MMTT in Efficacy Population 1
Description: C-peptide levels not normalized by the number of islet equivalent (IEQ)/kg were measured at the baseline in fasting condition, and at the following timepoints: 15, 30, 60, 90, 120 min after mixed meal at the hereunder reported time frame.
Time Frame: Day 75±5 after the 1st and 2nd islet infusion and day 365±14 after last islet infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
ng/mL
  Basal - day 75 - Transplant 1 | 0.50 (0.46) | 0.51 (0.44)
  15 min - day 75 - Transplant 1: number analyzed (Participants) | 26 | 18
  15 min - day 75 - Transplant 1 | 0.71 (0.77) | 0.67 (0.71)
  30 min - day 75 - Transplant 1: number analyzed (Participants) | 26 | 18
  30 min - day 75 - Transplant 1 | 1.18 (1.32) | 0.89 (0.90)
  60 min - day 75 - Transplant 1 | 1.66 (1.80) | 1.46 (1.43)
  90 min - day 75 - Transplant 1 | 1.81 (1.64) | 1.80 (1.57)
  120 min - day 75 - Transplant 1: number analyzed (Participants) | 27 | 17
  120 min - day 75 - Transplant 1 | 1.72 (1.34) | 2.04 (1.64)
  Basal - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  Basal - day 75 - Transplant 2 | 0.93 (0.69) | 1.27 (0.50)
  15 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  15 min - day 75 - Transplant 2 | 1.42 (1.36) | 1.73 (0.78)
  30 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  30 min - day 75 - Transplant 2 | 2.13 (1.90) | 2.55 (1.19)
  60 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  60 min - day 75 - Transplant 2 | 2.98 (2.15) | 3.65 (2.09)
  90 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  90 min - day 75 - Transplant 2 | 3.30 (2.15) | 3.56 (1.96)
  120 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  120 min - day 75 - Transplant 2 | 3.33 (1.98) | 2.90 (1.28)
  Basal - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  Basal - day 365 - Last transplant | 0.76 (0.65) | 1.14 (0.62)
  15 min - day 365 - Last transplant: number analyzed (Participants) | 23 | 15
  15 min - day 365 - Last transplant | 1.06 (1.02) | 1.32 (0.90)
  30 min - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  30 min - day 365 - Last transplant | 1.65 (1.66) | 2.17 (1.50)
  60 min - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  60 min - day 365 - Last transplant | 2.37 (2.38) | 2.88 (181)
  90 min - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  90 min - day 365 - Last transplant | 2.47 (2.27) | 3.13 (1.84)
  120 min - day 365 - Transplant 2: number analyzed (Participants) | 24 | 14
  120 min - day 365 - Transplant 2 | 2.11 (1.74) | 3.12 (1.68)

14. Secondary Outcome: Basal (Fasting) and 0 to 120 Min Time Course of Insulin Derived From the MMTT in Efficacy Population 1
Description: Insulin levels were measured at the baseline in fasting condition, and at the following timepoints: 15, 30, 60, 90, 120 min after mixed meal at the hereunder reported time frame.
Time Frame: Day 75±5 after the 1st and 2nd islet infusion and day 365±14 after last islet infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µU/mL
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
µU/mL
  Basal - day 75 - Transplant 1 | 16.5 (43.6) | 15.2 (39.8)
  15 min - day 75 - Transplant 1: number analyzed (Participants) | 23 | 17
  15 min - day 75 - Transplant 1 | 13.5 (16.6) | 11.8 (13.2)
  30 min - day 75 - Transplant 1: number analyzed (Participants) | 24 | 17
  30 min - day 75 - Transplant 1 | 21.0 (27.7) | 15.8 (16.9)
  60 min - day 75 - Transplant 1: number analyzed (Participants) | 25 | 17
  60 min - day 75 - Transplant 1 | 25.6 (32.9) | 23.0 (24.4)
  90 min - day 75 - Transplant 1: number analyzed (Participants) | 25 | 17
  90 min - day 75 - Transplant 1 | 23.9 (27.4) | 22.3 (18.8)
  120 min - day 75 - Transplant 1: number analyzed (Participants) | 25 | 16
  120 min - day 75 - Transplant 1 | 21.3 (28.2) | 23.1 (18.1)
  Basal - day 75 - Transplant 2: number analyzed (Participants) | 16 | 12
  Basal - day 75 - Transplant 2 | 8.4 (10.3) | 9.0 (3.8)
  15 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 11
  15 min - day 75 - Transplant 2 | 16.0 (16.0) | 17.5 (12.1)
  30 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 11
  30 min - day 75 - Transplant 2 | 28.4 (30.0) | 31.1 (17.8)
  60 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 11
  60 min - day 75 - Transplant 2 | 33.7 (23.4) | 37.8 (20.4)
  90 min - day 75 - Transplant 2: number analyzed (Participants) | 16 | 11
  90 min - day 75 - Transplant 2 | 36.3 (23.6) | 31.2 (20.6)
  120 min - day 75 - Transplant 2: number analyzed (Participants) | 17 | 11
  120 min - day 75 - Transplant 2 | 29.7 (19.2) | 25.3 (10.4)
  Basal - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  Basal - day 365 - Last transplant | 7.5 (7.6) | 6.2 (4.0)
  15 min - day 365 - Last transplant: number analyzed (Participants) | 23 | 15
  15 min - day 365 - Last transplant | 13.8 (17.0) | 10.8 (9.0)
  30 min - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  30 min - day 365 - Last transplant | 19.4 (19.2) | 20.7 (13.1)
  60 min - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  60 min - day 365 - Last transplant | 28.5 (30.1) | 25.6 (14.3)
  90 min - day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  90 min - day 365 - Last transplant | 25.8 (23.5) | 26.1 (17.8)
  120 min - day 365 - Transplant 2: number analyzed (Participants) | 24 | 14
  120 min - day 365 - Transplant 2 | 19.9 (18.4) | 27.1 (11.8)

15. Secondary Outcome: β-cell Function as Assessed by β-score in Efficacy Population 1
Description: The β-score ranges from 0 (no graft function) to 8 (interpreted as an index of excellent graft function), and gives 0-2 points each for glucose, HbA1C, stimulated C-peptide and insulin requirement. Both for the total and partial scores the higher the score, the better the outcome.
  Fasting plasma glucose (mg/dL): ≤99 (Score 2); 100 - 124 (Score 1); ≥125 (Score 0); HbA1c (%): ≤6.1(Score 2); 6.2 - 6.9 (Score 1); ≥ 7.0 (Score 0); Daily average (previous week) insulin (IU/kg/day): --- (Score 2); 0.01 - 0.24 (score 1); ≥ 0.25 (Score 0) Stimulated C-peptide (ng/mL): ≥ 0.9; 0.3 - 0.89; ≤0.3
Time Frame: Day 75±5 after the 1st and 2nd islet infusion and day 365±14 after last islet infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
score on a scale
  day 75 - Transplant 1 | 4.19 (2.37) | 4.06 (2.29)
  day 75 - Transplant 2: number analyzed (Participants) | 17 | 12
  day 75 - Transplant 2 | 5.53 (1.42) | 5.67 (2.06)
  day 365 - Last transplant: number analyzed (Participants) | 24 | 15
  day 365 - Last transplant | 4.63 (2.50) | 5.13 (2.42)
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; This is the analytic statistics for Day 75 (Transplant 1); Test type: Superiority; p = 0.9949, ANOVA — Treatment p value; Least square mean difference = 0.00, 95% CI 2-sided [-1.28 to 1.28]
Statistical Analysis 2: Comparison: Reparixin Group vs Placebo Group; This is the analytic statistics for Day 75 (Transplant 2); Test type: Superiority; p = 0.8753, ANOVA — Treatment p value; Least square mean difference = 0.10, 95% CI 2-sided [-1.18 to 1.38]
Statistical Analysis 3: Comparison: Reparixin Group vs Placebo Group; This is the analytic statistics for Day 365 (last Transplant); Test type: Superiority; p = 0.3955, ANOVA — Treatment p value; Least square mean difference = -0.59, 95% CI 2-sided [-1.97 to 0.80]

16. Secondary Outcome: β-cell Function as Assessed by Transplant Estimated Function (TEF) in Efficacy Population 1
Description: TEF selects the two pivotal components of the β-score (DIR and A1C) and links them together through a simple description of how insulin supply influences the patient's glycemic control.
  TEF was evaluated by the following equation: TEF = a.DIR + b.HbA1c + c where DIR = daily insulin requirement (average in the previous week); a = -1; b = 1/-5.43; c = -a.DIR (pre-transplant) - b.HbA1c (pre-transplant)
Time Frame: Day 75±5 after the 1st and 2nd islet infusion and day 365±14 after last islet infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/kg/24 h
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
U/kg/24 h
  day 75 - Transplant 1 | 0.523 (0.260) | 0.621 (0.332)
  day 75 - Transplant 2: number analyzed (Participants) | 18 | 15
  day 75 - Transplant 2 | 0.764 (0.240) | 0.981 (0.275)
  day 365 - Last transplant: number analyzed (Participants) | 25 | 16
  day 365 - Last transplant | 0.539 (0.320) | 0.719 (0.359)
Statistical Analysis 1: Comparison: Reparixin Group vs Placebo Group; This is the analytic statistics for Day 75 (Transplant 1); Test type: Superiority; p = 0.2444, ANOVA — Treatment p value; Least square mean difference = -0.105, 95% CI 2-sided [-0.286 to 0.075]
Statistical Analysis 2: Comparison: Reparixin Group vs Placebo Group; This is the analytic statistics for Day 75 (Transplant 2); Test type: Superiority; p = 0.0328, ANOVA — Treatment p value; Least square mean difference = -0.218, 95% CI 2-sided [-0.417 to -0.019]
Statistical Analysis 3: Comparison: Reparixin Group vs Placebo Group; This is the analytic statistics for Day 365 (last Transplant); Test type: Superiority; p = 0.1059, ANOVA — This is the analytic statistics for Day 75 (Transplant 2); Least square mean difference = -0.177, 95% CI 2-sided [-0.393 to 0.039]

17. Other Pre Specified Outcome: Frequency of Patients Positive/Negative for Autoantibodies Against Glutamic Acid Decarboxylase (GAD) in Efficacy Population 1
Description: Auto-antibodies were assayed on cell-free serum samples obtained as per centre practice ideally by immunoprecipitation of recombinant antigens. The Luminescent Immuno-Precipitation System based on chimeric autoantigens fused to luciferase enzyme was suggested as the preferred method to be used. Luciferase activity was measured in recovered immune-complex.
Time Frame: At pre-transplant, Day 75±5 after the 1st and 2nd islet infusion and Day 365±14 days after the last islet infusion
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
Percentage of participants
  pre-transplant 1 - positive: number analyzed (Participants) | 27 | 17
  pre-transplant 1 - positive | 48.1 | 52.9
  pre-transplant 1 - negative: number analyzed (Participants) | 27 | 17
  pre-transplant 1 - negative | 51.9 | 47.1
  day 75 - Transplant 1 - positive: number analyzed (Participants) | 26 | 17
  day 75 - Transplant 1 - positive | 69.2 | 64.7
  day 75 - Transplant 1 - negative: number analyzed (Participants) | 26 | 17
  day 75 - Transplant 1 - negative | 30.8 | 35.3
  pre-transplant 2 - positive: number analyzed (Participants) | 18 | 16
  pre-transplant 2 - positive | 66.7 | 62.5
  pre-transplant 2 - negative: number analyzed (Participants) | 18 | 16
  pre-transplant 2 - negative | 33.3 | 37.5
  day 75 - Transplant 2 - positive: number analyzed (Participants) | 18 | 15
  day 75 - Transplant 2 - positive | 66.7 | 53.3
  day 75 - Transplant 2 - negative: number analyzed (Participants) | 18 | 15
  day 75 - Transplant 2 - negative | 33.3 | 46.7
  day 365 - Last transplant - positive: number analyzed (Participants) | 25 | 16
  day 365 - Last transplant - positive | 56.0 | 50.0
  day 365 - Last transplant - negative: number analyzed (Participants) | 25 | 16
  day 365 - Last transplant - negative | 44.0 | 50.0

18. Other Pre Specified Outcome: Frequency of Patients Positive/Negative for Autoantibodies Against Islet Antigen-2 (IA-2) in Efficacy Population 1
Description: as for outcome 17
Time Frame: At pre-transplant, Day 75±5 after the 1st and 2nd islet infusion and Day 365±14 days after the last islet infusion,
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
Percentage of participants
  pre-transplant 1 - positive: number analyzed (Participants) | 27 | 14
  pre-transplant 1 - positive | 22.2 | 14.3
  pre-transplant 1 - negative: number analyzed (Participants) | 27 | 14
  pre-transplant 1 - negative | 77.8 | 85.7
  day 75 - Transplant 1 - positive: number analyzed (Participants) | 25 | 15
  day 75 - Transplant 1 - positive | 28.0 | 20.0
  day 75 - Transplant 1 - negative: number analyzed (Participants) | 25 | 15
  day 75 - Transplant 1 - negative | 72.0 | 80.0
  pre-transplant 2 - positive: number analyzed (Participants) | 18 | 15
  pre-transplant 2 - positive | 22.2 | 13.3
  pre-transplant 2 - negative: number analyzed (Participants) | 18 | 15
  pre-transplant 2 - negative | 77.8 | 86.7
  day 75 - Transplant 2 - positive: number analyzed (Participants) | 18 | 14
  day 75 - Transplant 2 - positive | 27.8 | 14.3
  day 75 - Transplant 2 - negative: number analyzed (Participants) | 18 | 14
  day 75 - Transplant 2 - negative | 72.2 | 85.7
  day 365 - Last transplant - positive: number analyzed (Participants) | 25 | 15
  day 365 - Last transplant - positive | 20.0 | 20.0
  day 365 - Last transplant - negative: number analyzed (Participants) | 25 | 15
  day 365 - Last transplant - negative | 80.0 | 80.0

19. Other Pre Specified Outcome: Frequency of Patients Positive/Negative for Autoantibodies Against Class I Human Leucocyte Antigen (HLA) in Efficacy Population 1
Description: Anti-HLA antibodies were assayed on cell-free serum samples obtained as per centre practice ideally by the Luminex analyzer. Class I and II positive/negative results were recorded.
Time Frame: Pre-transplant, day 75±5 after the 1st and 2nd islet infusion and day 365±14 after the last islet infusion
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
Percentage of participants
  pre-transplant 1 - positive | 15.4 | 27.8
  pre-transplant 1 - negative | 84.6 | 72.2
  day 75 - Transplant 1 - positive | 20.0 | 23.5
  day 75 - Transplant 1 - negative | 80.0 | 76.5
  pre-transplant 2 - positive | 29.4 | 31.3
  pre-transplant 2 - negative | 70.6 | 68.8
  day 75 - Transplant 2 - positive | 33.3 | 26.7
  day 75 - Transplant 2 - negative | 66.7 | 73.3
  day 365 - Last transplant - positive | 28.0 | 26.7
  day 365 - Last transplant - negative | 72.0 | 73.3

20. Other Pre Specified Outcome: Frequency of Patients Positive/Negative for Autoantibodies Against Class II Human Leucocyte Antigen (HLA) in Efficacy Population 1
Description: as for outcome 19
Time Frame: At pre-transplant, Day 75±5 after the 1st and 2nd islet infusion and Day 365±14 days after the last islet infusion,
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Reparixin Group | Placebo Group
Number analyzed (Participants) | 27 | 18
Percentage of participants
  pre-transplant 1 - positive | 7.7 | 5.6
  pre-transplant 1 - negative | 92.3 | 94.4
  day 75 - Transplant 1 - positive | 16.0 | 12.5
  day 75 - Transplant 1 - negative | 84.0 | 87.5
  pre-transplant 2 - positive | 5.9 | 6.3
  pre-transplant 2 - negative | 94.1 | 93.8
  day 75 - Transplant 2 - positive | 16.7 | 6.7
  day 75 - Transplant 2 - negative | 83.3 | 93.3
  day 365 - Last transplant - positive | 20.0 | 20.0
  day 365 - Last transplant - negative | 80.0 | 80.0

ADVERSE EVENTS:
Arm/Group | Reparixin Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/19
Serious Adverse Events (participants affected / at risk) | 17/29 | 12/19
Other Adverse Events (participants affected / at risk) | 29/29 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin Group (N=29) | Placebo Group (N=19)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intra-abdominal haemmorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (2)
Implant site haemorrhage (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hepatic haematoma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Alloimmunisation (Immune system disorders) | 2 (2) | 0 (0)
Drug Hypersensititity (Immune system disorders) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HLA marker study positive (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Panel-reactive antibody increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary retantion (Renal and urinary disorders) | 0 (0) | 1 (1)
Oropharyngeal ache (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin Group (N=29) | Placebo Group (N=19)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 2 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (3) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 7 (9)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 2 (3)
Lip oedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (17) | 12 (15)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 6 (6)
Catheter site haemorrhage (General disorders) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 3 (4) | 2 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Implant site haemorrhage (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 4 (5) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 6 (6)
Vessel puncture site erythema (General disorders) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (2) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural heamatoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 1 (2)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (2)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Portal vein presssure increased (Investigations) | 2 (2) | 1 (1)
Weight increased (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3)
joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (11) | 7 (9)
Migrane (Nervous system disorders) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (4)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin esfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No